CLINICAL TRIAL: NCT01552057
Title: A Phase III Clinical Trial of Duloxetine in Participants With Fibromyalgia
Brief Title: A Study of Duloxetine in Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14377; F1J-JE-HMGZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine 60 mg (Experimental): Duloxetine hydrochloride up to 60 milligrams (mg) orally for 15 weeks
  Interventions: Drug: Duloxetine 60 mg
- Placebo (Placebo Comparator): Placebo orally for 15 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine 60 mg — Duloxetine 60 mg taken orally once every day for 15 weeks
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine 60 mg
Drug: Placebo — Placebo taken orally once every day for 15 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the effectiveness and safety of duloxetine in participants with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Participants fulfilling the following criteria in the American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia
* Participants with pain rated severity 4 or over by Brief Pain Inventory (BPI) - average pain severity item (Question 3)

Exclusion Criteria:

* Participants with serious cardiovascular, hepatic, renal, respiratory, or hematological disease, or clinically significant laboratory or electrocardiogram abnormality which indicate a serious medical problem or require significant intervention in the judgment of the investigators
* Participants with alanine aminotransferase/aspartate aminotransferase of not less than 100 international units per liter (IU/L) or total bilirubin of not less than 1.6 milligrams per deciliter (mg/dL)
* Participants with serum creatinine level of not less than 2.0 mg/dL, participant who has undergone kidney transplantation or hemodialysis
* Participants with pain difficult to discriminate from pain associated with fibromyalgia or disease which disturbs the assessment
* Participants with treatment-refractory fibromyalgia
* Participants with thyroidal dysfunction, excluding those assessed by the investigator that the disorder is controlled as appropriate by 3-month or longer drug therapy
* Participants with present or past history of rheumatoid arthritis, inflammatory arthritis, infectious arthritis, or auto immune disease rather than thyroid deficiency
* Participants with an axis I condition according to Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV), currently or within the past year, except for major depressive disorders
* Participants with a lifetime diagnosis of bipolar disorder or schizoaffective disorder; or any other disorder with psychotic symptoms - based on the clinical opinion of the investigator
* Participants with personality disorder or mental retardation
* Participants with uncontrolled angle closure glaucoma
* Participants with present or past history of uncontrolled seizures or convulsion disorders
* Participants with suicidal ideation within past 6 months, with suicidal attempt within past 1 year
* Participants answering "yes" to any of the questions about active suicidal ideation/intent/behaviors occurring within the past 6 months (Columbia Suicide Severity Rating Scale, Suicide Ideation section - Questions 4 and 5; Suicidal Behavior section)
* Participants with past history of multiple episodes of drug allergy
* Female participants who are pregnant, lactating, or who want to get pregnant during the study period. Male participants who want his partner to get pregnant
* Females of child-bearing potential who can't agree to utilize medically. acceptable and reliable means of birth control during the study and for 1 month following the last dose of the study
* Participants with a history of alcohol or any psychoactive substance abuse or dependence (including alcohol, but excluding nicotine and caffeine) within the past 1 year
* Participants who have a positive urine drug screen for any substance of abuse (phencyclidine, cocaine, antihypnotic agent, or cannabis)
* Participants previously treated with duloxetine

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi, Japan

REFERENCES:
- [Derived] Murakami M, Osada K, Mizuno H, Ochiai T, Alev L, Nishioka K. A randomized, double-blind, placebo-controlled phase III trial of duloxetine in Japanese fibromyalgia patients. Arthritis Res Ther. 2015 Aug 22;17(1):224. doi: 10.1186/s13075-015-0718-y. PMID 26296539

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomized participants who completed the 14-week treatment period were considered to have completed the study. After study completion or early discontinuation, participants completed a 1-week taper and were observed 1 week post-treatment for safety.
Groups:
- Duloxetine 60 mg: Treatment Period: Up to 60-milligram (mg) dose of duloxetine administered orally once daily for 14 weeks. During the first 2 weeks of treatment, participants gradually increased their dosage. Week 1: 20-mg dose of duloxetine (one 20-mg capsule, and 2 placebo capsules), Week 2: 40-mg dose of duloxetine (two 20-mg capsules and 1 placebo capsule), Weeks 3 to 14: 60-mg dose of duloxetine (three 20-mg capsules).
  During the 1-week taper, the daily dosage was gradually reduced. For the first 3 days: 40-mg dose of duloxetine (two 20-mg capsules) administered orally once daily. For the remaining 4 days: 20-mg dose of duloxetine (one 20-mg capsule) administered orally once daily.
- Placebo: Treatment Period: 3 placebo capsules administered orally once daily for 14 weeks.
  During the 1-week taper, the number of placebo capsules was gradually reduced. For the first 3 days: 2 placebo capsules administered orally once daily. For the remaining 4 days: 1 placebo capsule administered orally once daily.
Period: Overall Study
Arm/Group | Duloxetine 60 mg | Placebo
Started | 196 | 197
Received at Least 1 Dose of Study Drug | 194 | 196
Completed | 166 | 149
Not Completed | 30 | 48
Not completed — Adverse Event | 14 | 15
Not completed — Lack of Efficacy | 8 | 23
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Entry Criteria Not Met | 2 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants who received at least 1 dose of study drug who had at least 1 post-baseline measurement of primary efficacy [Brief Pain Inventory (BPI) 24-hour average pain severity].
Groups:
- Duloxetine 60 mg: Treatment Period: Up to 60-mg dose of duloxetine administered orally once daily for 14 weeks. During the first 2 weeks of treatment, participants gradually increased their dosage. Week 1: 20-mg dose of duloxetine (one 20-mg capsule, and 2 placebo capsules), Week 2: 40-mg dose of duloxetine (two 20-mg capsules and 1 placebo capsule), Weeks 3 to 14: 60-mg dose of duloxetine (three 20-mg capsules).
  During the 1-week taper, the daily dosage was gradually reduced. For the first 3 days: 40-mg dose of duloxetine (two 20-mg capsules) administered orally once daily. For the remaining 4 days: 20-mg dose of duloxetine (one 20-mg capsule) administered orally once daily.
- Total: Total of all reporting groups
Arm/Group | Duloxetine 60 mg | Placebo | Total
Number analyzed (Participants) | 191 | 195 | 386
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (12.0) | 49.5 (11.7) | 48.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 164 | 321
  Male | 34 | 31 | 65
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 191 | 195 | 386
Region of Enrollment [Number; unit: participants]
  Japan | 191 | 195 | 386

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 14-Week Endpoint in the BPI 24-Hour Average Pain Severity Item of the BPI-Modified Short Form Score (MMRM)
Description: BPI 24-hour average pain severity is a self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. Severity scores ranged from 0 (no pain) to 10 (severe pain). Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach including administration groups, observation points, and interaction between the administration groups as fixed effects, and BPI average pain severity at baseline and the presence or absence of major depressive disorder as covariates; a linear model with unstructured error variance was applied.
Time Frame: Baseline, 14 weeks
Population: Randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline measurement of primary efficacy (BPI 24-hour average pain severity).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Duloxetine 60 mg: Treatment Period: Up to 60-mg dose of duloxetine administered orally once daily for 14 weeks. During the first 2 weeks of treatment, participants gradually increased their dosage. Week 1: 20-mg dose of duloxetine (one 20-mg capsule, and 2 placebo capsules), Week 2: 40-mg dose of duloxetine (two 20-mg capsules and 1 placebo capsule), Weeks 3 to 14: 60-mg dose of duloxetine (three 20-mg capsules).
- Placebo: Treatment Period: 3 placebo capsules administered orally once daily for 14 weeks.
Arm/Group | Duloxetine 60 mg | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale | -1.90 (0.23) | -1.58 (0.23)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.0988, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.70 to 0.06]

2. Secondary Outcome: Patients Global Impression of Improvement (PGI-I) at Endpoint
Description: PGI-I measures the participant's perception of improvement at the time of assessment compared with the start of treatment. Scores ranged from 1 (very much better) to 7 (very much worse). LS mean was calculated using an MMRM approach including administration groups, observation points, and interaction between the administration groups as fixed effects, and the presence or absence of major depressive disorder as covariates; a linear model with unstructured error variance was applied.
Time Frame: 14 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale | 2.83 (0.16) | 3.32 (0.16)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.0003, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.76 to -0.22]

3. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) at Endpoint
Description: CGI-I measures the clinician's perception of participant improvement at the time of assessment (compared with the start of treatment). Scores ranged from 1 (very much better) to 7 (very much worse). LS mean was calculated using an MMRM approach including administration groups, observation points, and interaction between the administration groups as fixed effects, and the presence or absence of major depressive disorder as covariates; a linear model with unstructured error variance was applied.
Time Frame: 14 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale | 2.83 (0.15) | 3.27 (0.16)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; p = 0.0012, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.71 to -0.18]

4. Secondary Outcome: Change From Baseline to 14-Week Endpoint in Fibromyalgia Impact Questionnaire (FIQ)
Description: FIQ is a 20-item, self-administered questionnaire using Likert-type scales to measure participant (pt) outcomes over the past week. Items 1 through 11 measured physical functioning on 4-point scales. Items 12 and 13 measured the number of days a pt felt well and days a pt was unable to work due to fibromyalgia symptoms. Items 14 through 20 were 11-point scales on which a pt rated work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety, and depression. If a pt did not do all the tasks listed, those items were deleted from scoring. Algorithms were used to determine total FIQ scores which ranged from 0 to 100; higher scores indicated a more negative impact. LS mean was calculated using an MMRM approach including administration groups, observation points, and interaction between administration groups as fixed effects, and baseline as well as the presence or absence of major depressive disorder as covariates; a linear model with unstructured error variance was applied.
Time Frame: Baseline, 14 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale | -18.41 (2.57) | -13.05 (2.65)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.0073, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -5.35, 95% CI 2-sided [-9.26 to -1.45]

5. Secondary Outcome: Change From Baseline to 14-Week Endpoint in 36-Item Short-Form (SF-36) Health Survey Domain Scores
Description: The SF-36 Health Survey is a generic, health-related survey assessing the participant's quality of life on 8 domains: physical functioning, daily functioning (physical), bodily pain, general health, vitality, social functioning, daily functioning (emotional), and mental health. Each domain was scored by summing individual items pertaining to that domain and transforming scores into a 0 to 100 scale, with higher scores indicating better health status or functioning. LS mean was calculated using an ANCOVA approach including administration groups as fixed effects, and baseline as well as the presence or absence of complication by major depressive disorder as covariates.
Time Frame: Baseline, up to 14 weeks
Population: Randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline measurement of primary efficacy (BPI 24-hour average pain severity); LOCF values were used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale
  Physical Functioning | 7.40 (2.13) | 3.06 (2.15)
  Role-Physical | 8.20 (2.96) | 0.44 (2.98)
  Bodily Pain | 10.95 (2.07) | 5.28 (2.08)
  General Health | 6.55 (1.92) | 3.31 (1.94)
  Vitality | 10.05 (2.51) | 3.35 (2.53)
  Social Functioning | 10.32 (3.04) | 3.28 (3.06)
  Role-Emotional | 5.50 (3.35) | -3.63 (3.36)
  Mental Health | 5.91 (2.51) | -2.00 (2.52)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; Physical Functioning; Test type: Superiority or Other; p = 0.0049, ANCOVA — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = 4.34, 95% CI 2-sided [1.32 to 7.35]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Role-Physical; Test type: Superiority or Other; p = 0.0003, ANCOVA — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = 7.76, 95% CI 2-sided [3.57 to 11.94]
Statistical Analysis 3: Comparison: Duloxetine 60 mg vs Placebo; Bodily Pain; Test type: Superiority or Other; p = 0.0002, ANCOVA — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = 5.67, 95% CI 2-sided [2.76 to 8.59]
Statistical Analysis 4: Comparison: Duloxetine 60 mg vs Placebo; General Health; Test type: Superiority or Other; p = 0.0192, ANCOVA — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = 3.25, 95% CI 2-sided [0.53 to 5.96]
Statistical Analysis 5: Comparison: Duloxetine 60 mg vs Placebo; Vitality; Test type: Superiority or Other; p = 0.0002, ANCOVA — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = 6.70, 95% CI 2-sided [3.15 to 10.25]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Placebo; Social Functioning; Test type: Superiority or Other; p = 0.0014, ANCOVA — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = 7.04, 95% CI 2-sided [2.74 to 11.34]
Statistical Analysis 7: Comparison: Duloxetine 60 mg vs Placebo; Role-Emotional; Test type: Superiority or Other; p = 0.0002, ANCOVA — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = 9.12, 95% CI 2-sided [4.41 to 13.83]
Statistical Analysis 8: Comparison: Duloxetine 60 mg vs Placebo; Mental Health; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = 7.91, 95% CI 2-sided [4.39 to 11.43]

6. Secondary Outcome: Change From Baseline to 14-Week Endpoint in Beck Depression Inventory-II (BDI-II)
Description: The BDI-II is a 21-item self-administered questionnaire designed to assess the characteristics of depression. Each item was scored on a 4-point scale ranging from 0 (not present) to 3 (present in the extreme) and was summed to give a total BDI-II score. A total BDI-II score of 0 through 13 was considered minimal, 14 through 19 was mild, 20 through 28 was moderate, and 29 through 63 was severe depression symptoms. LS mean was calculated using an MMRM approach including administration groups, observation points, and interaction between the administration groups and as fixed effects, and baseline as well as the presence or absence of major depressive disorder as covariates; a linear model with unstructured error variance was applied.
Time Frame: Baseline, 14 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale | -4.07 (0.84) | -1.22 (0.85)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.0002, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -2.85, 95% CI 2-sided [-4.32 to -1.38]

7. Secondary Outcome: Change From Baseline to 14-Week Endpoint in Widespread Pain Index (WPI) and Symptom Severity (SS) in American College of Rheumatology (ACR) Fibromyalgia Diagnostic Criteria 2010
Description: WPI: Participant-reported areas (out of 19 points on the body) in which the participant had pain in the past week. WPI scores ranged from 0 (no areas) to 19 (all areas). SS: The sum of severity scores for fatigue, waking unrefreshed, and cognitive symptoms [each rated from 0 (no problem) to 3 (severe; life-disturbing problems)] plus the severity of somatic symptoms in general [rated from 0 (no symptoms) to 3 (a great deal of symptoms)]. The total SS score ranged from 0 and 12. LS mean was calculated using an MMRM approach including administration groups, observation points, interaction between the administration groups and the observation points as fixed effects, and baseline as well as the presence or absence of major depressive disorder as covariates; a linear model with unstructured error variance was applied.
Time Frame: Baseline, 14 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale
  WPI | -2.34 (0.58) | -1.06 (0.60)
  SS | -1.37 (0.27) | -1.00 (0.28)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; WPI; Test type: Superiority or Other; p = 0.0029, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-2.12 to -0.44]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Symptom Severity; Test type: Superiority or Other; p = 0.0906, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.79 to 0.06]

8. Secondary Outcome: Change From Baseline to 14-Week Endpoint in Average Pain and Worst Pain Severity Score Within 24-Hours in Participant Diary
Description: Each morning participants rated their average pain and worst pain within the past 24 hours on separate 11-point Likert scales with scores ranging from 0 (no pain) through 10 (worst possible pain). These scores were then averaged for the week and compared to baseline. LS mean was calculated using an MMRM approach including administration groups, observation points, and interaction between the administration groups as fixed effects, and baseline as well as the presence or absence of major depressive disorder as covariates; a linear model with unstructured error variance was applied.
Time Frame: Baseline, 14 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale
  Average Pain | -1.82 (0.18) | -1.48 (0.18)
  Worst Pain | -1.81 (0.19) | -1.34 (0.19)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; Average Pain; Test type: Superiority or Other; p = 0.0755, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.70 to 0.03]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Worst Pain; Test type: Superiority or Other; p = 0.0232, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.88 to -0.06]

9. Secondary Outcome: Change From Baseline to 14-Week Endpoint in Brief Pain Inventory-Severity (BPI-S) and Brief Pain Inventory-Interference (BPI-I) Scores on the BPI-Modified Short Form
Description: BPI-S and BPI-I are self-reported scales measuring severity of pain and interference on function, respectively. Severity scores ranged from 0 (no pain) to 10 (severe pain) for each question assessing worst pain, least pain, and pain right now. Interference scores ranged from 0 (does not interfere) to 10 (completely interferes) for each question assessing interference of pain in past 24 hours with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference was the average of non-missing scores of individual interference items. LS mean was calculated using an MMRM approach including administration groups, observation points, and interaction between the administration groups as fixed effects, and baseline as well as the presence or absence of major depressive disorder as covariates; a linear model with unstructured error variance was applied.
Time Frame: Baseline, 14 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale
  Worst Pain | -1.91 (0.26) | -1.35 (0.26)
  Least Pain | -1.72 (0.22) | -1.23 (0.22)
  Pain Right Now | -1.77 (0.26) | -1.20 (0.26)
  Interference With General Activity | -2.22 (0.31) | -1.76 (0.32)
  Interference With Mood | -2.17 (0.32) | -1.42 (0.33)
  Interference With Walking Ability | -1.67 (0.29) | -1.29 (0.30)
  Interference With Normal Work | -2.18 (0.31) | -1.76 (0.32)
  Interference With Relations With Other People | -1.09 (0.30) | -0.53 (0.30)
  Interference With Sleep | -1.82 (0.35) | -1.57 (0.36)
  Interference With Enjoyment of Life | -1.90 (0.31) | -1.24 (0.32)
  Average Interference | -1.95 (0.27) | -1.44 (0.27)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; Worst Pain; Test type: Superiority or Other; p = 0.0126, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-0.99 to -0.12]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Least Pain; Test type: Superiority or Other; p = 0.0092, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.87 to -0.12]
Statistical Analysis 3: Comparison: Duloxetine 60 mg vs Placebo; Pain Right Now; Test type: Superiority or Other; p = 0.0083, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.00 to -0.15]
Statistical Analysis 4: Comparison: Duloxetine 60 mg vs Placebo; Interference With General Activity; Test type: Superiority or Other; p = 0.0807, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.98 to 0.06]
Statistical Analysis 5: Comparison: Duloxetine 60 mg vs Placebo; Interference With Mood; Test type: Superiority or Other; p = 0.0057, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.29 to -0.22]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Placebo; Interference With Walking Ability; Test type: Superiority or Other; p = 0.1114, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.84 to 0.09]
Statistical Analysis 7: Comparison: Duloxetine 60 mg vs Placebo; Interference With Normal Work; Test type: Superiority or Other; p = 0.1081, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.94 to 0.09]
Statistical Analysis 8: Comparison: Duloxetine 60 mg vs Placebo; Interference With Relationships With Other People; Test type: Superiority or Other; p = 0.0264, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-1.04 to -0.07]
Statistical Analysis 9: Comparison: Duloxetine 60 mg vs Placebo; Interference With Sleep; Test type: Superiority or Other; p = 0.3959, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.81 to 0.32]
Statistical Analysis 10: Comparison: Duloxetine 60 mg vs Placebo; Interference With Enjoyment of Life; Test type: Superiority or Other; p = 0.0119, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-1.18 to -0.15]
Statistical Analysis 11: Comparison: Duloxetine 60 mg vs Placebo; Average Interference; Test type: Superiority or Other; p = 0.0222, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.96 to -0.07]

10. Primary Outcome: Change From Baseline to 2 Weeks in the BPI 24-Hour Average Pain Severity Item of the BPI-Modified Short Form Score (MMRM)
Description: BPI 24-hour average pain severity is a self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. Severity scores ranged from 0 (no pain) to 10 (severe pain). LS mean was calculated using an MMRM approach including administration groups, observation points, and interaction between the administration groups as fixed effects, and BPI average pain severity at baseline and the presence or absence of major depressive disorder as covariates; a linear model with unstructured error variance was applied.
Time Frame: Baseline, 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale | -1.00 (0.21) | -0.60 (0.22)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.0113, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.71 to -0.09]

11. Primary Outcome: Change From Baseline to 4 Weeks in the BPI 24-Hour Average Pain Severity Item of the BPI-Modified Short Form Score (MMRM)
Description: as for outcome 10
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale | -1.55 (0.22) | -0.94 (0.22)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.0005, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.94 to -0.27]

12. Primary Outcome: Change From Baseline to 6 Weeks in the BPI 24-Hour Average Pain Severity Item of the BPI-Modified Short Form Score (MMRM)
Description: as for outcome 10
Time Frame: Baseline, 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale | -1.81 (0.22) | -1.09 (0.23)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-1.07 to -0.37]

13. Primary Outcome: Change From Baseline to 10 Weeks in the BPI 24-Hour Average Pain Severity Item of the BPI-Modified Short Form Score (MMRM)
Description: as for outcome 10
Time Frame: Baseline, 10 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale | -1.85 (0.23) | -1.41 (0.23)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.0226, MMRM — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.82 to -0.06]

14. Primary Outcome: Change From Baseline up to 14-Week Endpoint in the BPI 24-Hour Average Pain Severity Item of the BPI-Modified Short Form Score (ANCOVA)
Description: BPI 24-hour average pain severity is a self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. Severity scores ranged from 0 (no pain) to 10 (severe pain). LS mean was calculated using an analysis of covariance (ANCOVA) approach including administration groups as fixed effects, and BPI average pain severity at baseline and the presence or absence of major depressive disorder as covariates.
Time Frame: Baseline, up to 14 weeks
Population: Randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline measurement of primary efficacy (BPI 24-hour average pain severity); Last Observation Carried Forward (LOCF) values were used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale | -1.60 (0.26) | -1.22 (0.26)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.0408, ANCOVA — Statistical tests were conducted at a 2-sided alpha level of 0.05; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.74 to -0.02]

ADVERSE EVENTS:
Time Frame: Baseline through 1 week post last dose
Description: Randomized who received at least 1 dose of study drug.
Arm/Group | Duloxetine 60 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/194 | 1/196
Other Adverse Events (participants affected / at risk) | 147/194 | 122/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine 60 mg (N=194) | Placebo (N=196)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Duloxetine 60 mg (N=194) | Placebo (N=196)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 5 (5) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 5 (6) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6) | 4 (4)
Constipation (Gastrointestinal disorders) | 29 (29) | 8 (8)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 7 (8)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 42 (44) | 9 (9)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (5) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7) | 4 (4)
Asthenia (General disorders) | 4 (4) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 2 (3) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 9 (9) | 6 (6)
Oedema (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Thirst (General disorders) | 14 (14) | 7 (7)
Hepatic function abnormal (Hepatobiliary disorders) | 5 (5) | 4 (4)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 3 (4) | 3 (3)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Keratitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 26 (39) | 29 (37)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Pertussis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heat illness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 5 (6) | 4 (4)
Blood cholesterol increased (Investigations) | 2 (2) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 3 (3)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 2 (2) | 2 (2)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 4 (4) | 4 (4)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Haematocrit increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 1 (1) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Red blood cell count increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (1)
Weight increased (Investigations) | 1 (1) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 13 (13) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypouricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 11 (11) | 2 (2)
Dizziness postural (Nervous system disorders) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 9 (11) | 6 (6)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 2 (2)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Sleep paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 51 (52) | 21 (21)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 5 (5)
Limited symptom panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Middle insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0/35 (0) | 1/31 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 1/159 (1) | 0/165 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1/159 (1) | 0/165 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Yawning (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 8 (8)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days